CLINICAL TRIAL: NCT02932839
Title: Investigating the Neuronal Bases of Epilepsy With Micro-electrode Arrays in Patients Who Are Candidates for Epilepsy Surgery
Brief Title: Investigating the Neuronal Bases of Epilepsy With Micro-electrode Arrays in Candidates for Epilepsy Surgery
Acronym: IN-MAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyss Center for Bio and Neuroengineering (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IN-MAP
Record Dates: First submitted 2016-09-26; First posted 2016-10-13 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-03

CONDITIONS: Epilepsy
Keywords: Epilepsy surgery; Micro-electrode arrays; Single-neuron recordings; Electrocorticography
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Implantation of the Blackrock NeuroPort micro-electrode array for up to 29 days in patients who are undergoing evaluation with intracranial EEG electrodes
  Interventions: Device: NeuroPort micro-electrode array

INTERVENTIONS:
Device: NeuroPort micro-electrode array — Implantation of the Blackrock NeuroPort micro-electrode array for up to 29 days in patients who are undergoing evaluation with intracranial EEG electrodes
  Other Names: Blackrock Microsystems

SUMMARY:
This study aims to uncover the neuronal bases of epilepsy by recording the activity of single neurons in the brain of patients with epilepsy who are candidates for assessment with intracranial electroencephalography (EEG). A micro-electrode array will be inserted into the brain in addition to the standard intracranial EEG electrodes for up to 4 weeks.

DETAILED DESCRIPTION:
Epilepsy is a disease characterized by the tendency to have seizures, which are thought to be due to excessive activity in the neurons of the brain. However, it is technically difficult to record the activity of neurons, especially in the brain of human patients. Therefore, there are gaps in what scientists know of what exactly goes wrong in neurons during epileptic seizures.

In this study, an array of micro-electrodes will be inserted into the brain of patients with epilepsy while they are undergoing a clinically indicated assessment with intracranial electroencephalography (EEG). The micro-electrode array is able to continuously record the activity of neurons in the human brain. In combination with the standard intracranial EEG, the recordings of the micro-electrode array will allow a better understanding of the relationship between epileptic seizures and the activity of neurons.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years old or older
* Patient who suffers from potentially surgically remediable drug-resistant focal epilepsy
* Patient in whom neocortical resective surgery is deemed likely
* Patient who requires evaluation with intracranial subdural EEG electrodes
* Patient in whom a cortical area that is not eloquent (i.e. not involved in a critical neurological function like language or motor control) is deemed highly likely to be involved in seizure onset or propagation and is therefore an appropriate site for the implantation of the micro-electrode array
* Patient who is able and willing to provide informed consent

Exclusion Criteria:

* Patient in whom neocortical resective surgery is deemed unlikely (e.g. patients in whom a corpus callosotomy or another palliative epilepsy surgery procedure is planned)
* Patient who will be investigated with stereo-EEG electrodes only (these patients will not undergo a craniotomy for clinical purposes, and implantation of the micro-electrode array is therefore impossible)
* Patient whose epileptic seizures cause hypermotor or violent motor behavior (due to the risk of MD mechanical failure and related injury)
* Patient with a previous history of bacterial meningitis (due to the risk of thickening of the arachnoid membrane complicating the implantation of the micro-electrode array)
* Patient with severe psychiatric disease or psychological distress
* Patient with severe concomitant medical disease (including, but not limited to, cardiovascular disease, respiratory illness, renal failure, hepatic dysfunction, etc.)
* Patient with known compromise of the immune system caused by a medical condition or the chronic consumption of immunosuppressant medication (due to the increased risk of infection; this includes diabetes mellitus)
* Patient with colonization with methicillin-resistant Staphylococcus aureus (due to the increased risk of difficult-to-manage infection)
* Patient with known tendency for increased bleeding (due to the increased risk of hemorrhage)
* Patient with an implanted intracranial stimulator, vagus nerve stimulator, or cochlear implant that will remain active during the study (due to the potential for interference with the micro-electrode recordings)
* Women who are pregnant or breastfeeding during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with study procedure- and investigational device-related serious adverse events, as defined in ISO 14155 | On average 4 weeks
  Number of patients experiencing any serious adverse event, as defined in ISO 14155 (any untoward medical occurrence that resulted in death or led to a serious deterioration in health), that is possibly, probably or definitely related to study procedures or the investigational device. Participants will be hospitalized throughout the duration of their participation in the study. Serious adverse events will be monitored daily by a physician through history taking, neurological examination, measurements of vital signs as well as every other day with blood testing for markers of inflammation (leucocytosis and elevated C-reactive protein).
Correlation between EEG markers of epileptic activity and single-neuron activity recorded by the investigational device | Up to 4 weeks
  The characteristics of single-neuron activity (recorded by the investigational device) will be studied during epileptic events as identified by the clinical intracranial EEG (interictal epileptic discharges, high-frequency oscillations, epileptic seizures), including (not necessarily limited to) average firing rate, across-neuron firing synchronization, phase-amplitude coupling with slow cortical oscillations. These analyses will be performed using specialized, custom-programmed neural time series data processing software.

SECONDARY OUTCOMES:
Number of single neurons recorded from investigational device | Up to 4 weeks
  Number of single neurons isolated by the investigational device and stability over time of these recordings. These analyses will be performed using specialized, custom-programmed neural time series data processing software.

CONTACTS AND LOCATIONS:
Overall Officials: Margitta Seeck, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided